CLINICAL TRIAL: NCT02720913
Title: COR-KNOT Versus Manually Hand-tied Knots
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Marc Gillinov, MD, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-159
Record Dates: First submitted 2016-03-14; First posted 2016-03-28 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Suture Tying
Keywords: Time; COR-KNOT; Standard; Cost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COR-KNOT (Experimental): The COR-KNOT device was developed to make suture fixation faster and save operative time. With a single squeeze of the lever, the device remotely and automatically secures sutures with a titanium fastener, while also simultaneously trimming excess suture tails.
  Interventions: Device: COR-KNOT
- Standard Suture Tying (Active Comparator): Standard Suture Tying
  Interventions: Procedure: Standard Suture Tying

INTERVENTIONS:
Device: COR-KNOT — The COR-KNOT device was developed to make suture fixation faster and save operative time. With a single squeeze of the lever, the device remotely and automatically secures sutures with a titanium fastener, while also simultaneously trimming excess suture tails.
  Arms: COR-KNOT
Procedure: Standard Suture Tying — Standard Suture Tying
  Arms: Standard Suture Tying

SUMMARY:
The COR-KNOT technology (LSI SOLUTIONS, Victor, New York USA) was developed to replace suture tying with a faster procedure during surgery. While preclinical studies confirmed the speed of COR-KNOT use, no clinical studies have quantitatively compared the speed of suture fixation delivered by the COR-KNOT device with the speed of conventional hand-tied knots. COR-KNOT is expensive, costing 189 $ per application. Given this added expense, it is important to quantify the time-saved by application of this technology.

DETAILED DESCRIPTION:
The COR-KNOT device was developed to make suture fixation faster and save operative time. With a single squeeze of the lever, the device remotely and automatically secures sutures with a titanium fastener, while also simultaneously trimming excess suture tails. This device has been accepted by cardiac surgeons for the recognized benefits of time savings, simplicity, and reliability.

While the device presents ergonomic advantages during minimally invasive cardiac surgery, it enjoys widespread use in sternotomy-based, standard heart surgery. The relative cost of the device as a function of time saved has not been assessed. The purpose of this trial is to determine the relative time savings and cost of COR-KNOT compared to standard hand-tied knots in patients undergoing mitral/tricuspid ring annuloplasty repairs via traditional open heart surgery. Valve repair surgery is a common setting for COR-KNOT use and therefore serves as an appropriate procedure for evaluation of the technology.

The investigators propose a prospective, randomized trial in patients undergoing mitral or tricuspid ring annuloplasty repair to 1) Determine the time require per knot for COR-KNOT versus standard hand-tied knots and 2) Quantify the relative cost of COR-KNOT versus that of standard, hand-tied knots. Data from this study will enable the investigators to determine the cost-benefit of using COR-KNOT technology in cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for Valvular ring annuloplasty for mitral and/or tricuspid valve repair
* Age > 18 years
* Able and willing to give informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01-11 (Actual)

PRIMARY OUTCOMES:
Time (seconds) required to use COR-KNOT vs. Standard Suture Tying | 60 seconds

SECONDARY OUTCOMES:
Cost (US Dollar) of using COR-KNOT vs. Standard Suture Tying | 60 seconds
  Assess cost using manufacturer price quotes (US$)

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Gillinov, MD, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No